CLINICAL TRIAL: NCT00124137
Title: Ultrafiltration Versus IV Diuretics for Patients Hospitalized for Acute Decompensated Heart Failure: A Prospective Randomized Clinical Trial
Brief Title: Ultrafiltration Versus Intravenous (IV) Diuretics for Patients Hospitalized for Acute Decompensated Heart Failure: (UNLOAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuwellis, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-1
Record Dates: First submitted 2005-07-25; First posted 2005-07-27 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2005-12

CONDITIONS: Congestive Heart Failure
Keywords: Ultrafiltration; acute decompensated heart failure; fluid overload; pulmonary congestion
MeSH Terms: conditions — Heart Failure; Edema | interventions — Diuretics

INTERVENTIONS:
Device: Aquadex system
Drug: IV diuretic

SUMMARY:
The purpose of this study is to compare patients who are suffering from heart failure and who are fluid overloaded to determine if ultrafiltration (UF) can remove more of the extra fluid as measured by weight loss while in the hospital and improve the patient's breathing.

DETAILED DESCRIPTION:
Congestive heart failure is an important public health issue. It remains the leading cause of hospitalization in Medicare beneficiaries. Ninety percent of all hospitalizations for CHF are due to fluid overload. Most of the expense related to the management of heart failure is due to hospital-based care; interventions that reduce the amount of time patients spend in the hospital may greatly decrease the cost associated with caring for these patients.

Hospital stay for patients admitted for acute decompensated congestive heart failure (adCHF) is largely dictated by how quickly the signs and symptoms of congestion can be relieved and whether ACE inhibitors can be started safely. Diuretics are usually effective in relieving congestion, but achieving adequate diuresis often requires a process of trial and error. Some patients are simply refractory to oral or intravenous diuretics. Diuretics stimulate adverse neurohormonal systems and can cause progressive azotemia. Bayliss (1977) showed that there is a significant increase in renin and aldosterone levels as a response to diuretic treatment rather than as a result of the heart failure itself. Gottlieb (2002) showed that loop diuretics diminish glomerular filtration rate in patients with heart failure. In addition, as more diuretics are given, serum electrolyte imbalances often occur, requiring additional monitoring of patients.

UF has been used as a therapeutic method to remove excessive fluid in patients for over 30 years. UF removes excess water without causing a significant clinical change in the electrolyte composition of the blood or causes adverse affects on the kidneys and neurohormonal system. Studies have shown that UF increases urine output, increases responsiveness to standard oral therapies and decreases readmission rate. While the usefulness of UF in this patient population has great potential, this form of therapy is not usually performed due to the need for invasive venous access and increased expense i.e. high flow dialysis machines. CHF Solutions has developed the Aquadex System that has FDA market clearance for UF. The advantage of the Aquadex System is its simplicity and the fact that it can be administered by means of peripheral catheters or with a central venous access. Early prospective series and subsequent clinical experience involving adCHF patients have shown that 4 to 8 liters can easily be withdrawn in a short amount of time using the peripheral access approach with the Aquadex System. Volume removal was not associated with disruption of electrolyte balance, worsening of renal distress or impact on blood pressure or heart rate of clinical significance. The Aquadex System is a predictable, safe, and effective way to ensure adequate volume removal that may result in shorter hospital stays, better symptom relief and more efficient dosing of medications for the treatment of adCHF.

The purpose of this study is to determine whether the Aquadex System can improve the acute management of patients with adCHF and maintain this improvement over a period of time compared to IV diuretics. Ultrafiltration in this patient population may decrease length of hospital stay and reduce hospital readmissions for heart failure leading to a significant reduction in costs for the treatment of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with primary diagnosis of acute decompensated congestive heart failure (adCHF)
* Evidence of fluid overload as indicated by:

  1. pitting edema (2+) of lower extremities;
  2. jugular venous distension;
  3. pulmonary edema or pleural effusion;
  4. ascites;
  5. paroxysmal nocturnal dyspnea or 2-pillow orthopnea

Exclusion Criteria:

* Acute coronary syndrome
* Creatinine greater than 3.0
* Systolic blood pressure less than or equal to 90 mmHg
* Hematocrit greater than 45%
* Prior administration of IV vasoactive drugs in the emergency room (ER)
* Clinical instability requiring pressors during hospitalization
* Recent use of iodinated contrast material
* Severe concomitant disease expected to prolong hospitalization
* Sepsis
* On or requires renal dialysis
* Had a cardiac transplant
* Heparin allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-04; Study Completion 2005-10

PRIMARY OUTCOMES:
Total weight loss during first 48 hours of randomization
Change in dyspnea score during first 48 hours of randomization

SECONDARY OUTCOMES:
Change in global assessment
Change in quality of life (living with heart failure)
Changes in brain natriuretic peptide (BNP)
Changes in 6 minute walk test
Total fluid loss during first 48 hours of randomization
Changes in blood urea nitrogen (BUN) and creatinine
Changes in renin and aldosterone

CONTACTS AND LOCATIONS:
Overall Officials: Maria R Costanzo, MD, Principal Investigator — Midwest Heart
Locations (1):
- Midwest Heart Institute, Lombard, Illinois, United States

REFERENCES:
- [Derived] Costanzo MR, Guglin ME, Saltzberg MT, Jessup ML, Bart BA, Teerlink JR, Jaski BE, Fang JC, Feller ED, Haas GJ, Anderson AS, Schollmeyer MP, Sobotka PA; UNLOAD Trial Investigators. Ultrafiltration versus intravenous diuretics for patients hospitalized for acute decompensated heart failure. J Am Coll Cardiol. 2007 Feb 13;49(6):675-83. doi: 10.1016/j.jacc.2006.07.073. Epub 2007 Jan 26. PMID 17291932